CLINICAL TRIAL: NCT01079845
Title: Low-glycemic Load vs. Low-fat Diet for Treating PCOS in Obese Adolescents and Young Adults
Brief Title: A Cooking and Eating Study
Acronym: ACES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For this pilot, we constructed conditional power curves and noted that we would not substantially enhance power by enrolling additional participants.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Cara Ebbeling, Associate Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02-0069
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Diet; Nutrition; Adolescent; Young Adult; Overweight; Obesity
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight; Obesity | interventions — Nutrition Assessment; Cooking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-glycemic Load Diet (Experimental)
  Interventions: Behavioral: Nutrition Education, Dietary Counseling, and Cooking
- Low-fat Diet (Active Comparator)
  Interventions: Behavioral: Nutrition Education, Dietary Counseling, and Cooking

INTERVENTIONS:
Behavioral: Nutrition Education, Dietary Counseling, and Cooking — Monthly clinic visits with a dietitian, Monthly telephone calls with a dietitian, Three cooking workshops with a chef

SUMMARY:
Background. The polycystic ovary syndrome (PCOS) is a complex hormonal disorder that presents in susceptible girls around the time of menarche. Females with PCOS have high levels of androgens (e.g., testosterone). While cosmetic appearance (excess facial hair and acne) and menstrual disturbances were once considered the primary concerns, emerging data indicate that many adolescents and young adults with PCOS are insulin resistant and at increased risk for metabolic syndrome and diabetes. The majority of females with PCOS are obese, and excess body fat amplifies the severity of the syndrome.

Dietary intervention is considered an important component of treatment for PCOS. However, a consensus statement regarding optimal nutrient composition for treating adolescents and young adults with PCOS has not been published because data are lacking to provide a foundation for such a statement. Recognizing increased risk for diabetes in patients with PCOS, many practitioners employ a low-fat diet as prescribed in the Diabetes Prevention Program (DPP) for weight loss and control of symptoms.

Objective and Hypothesis. The purpose of this research study is to compare different diets for treating PCOS. We hypothesize that a low-glycemic load diet - designed to lower blood levels of glucose and insulin - will be more beneficial than a low-fat diet in obese adolescents and young adults with PCOS.

Design. We propose a 6-month study in which 50 obese females with PCOS (ages 13 to 21 years) will be assigned to receive one of two dietary treatments, with the goal of retaining 40 participants. Group assignment will be at random. One of the treatments will be a low-glycemic load diet, and the other treatment will be a low-fat diet (modeled after the DPP diet). Participants in both groups will receive individual nutrition education and dietary counseling with a registered dietitian (clinic visits, telephone calls) and cooking workshops with a chef. The purpose of the cooking workshops will be to enhance compliance with diet prescriptions, beyond what can be achieved by nutrition education and dietary counseling in a conventional clinic setting.

The primary outcome will be bioavailable testosterone (form of testosterone that causes symptoms of PCOS). Secondary outcomes will include other blood tests to evaluate further high androgen levels (total testosterone, free testosterone, sex hormone binding globulin, dehydroepiandrosterone sulfate), clinical signs of high androgen levels (excess facial hair, acne), glucose tolerance and risk for diabetes (determined by blood sugar and insulin measurements), risk for cardiovascular disease (based on blood cholesterol and C-reactive protein levels and blood pressure), body fat percentage and distribution (measured using state-of-the-art dual energy x-ray absorptiometry and waist circumference), menstrual cyclicity, and health-related quality of life (evaluated by questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS.
* Aged 13 to 21 years (and living at home with a parent, only for those <18 years old).
* Body mass index (BMI) at or above the 85th percentile.
* Access to a working telephone.
* At least one parent willing and able to participate in the intervention, only for those <18 years old.
* Residing in predominately one household (no more than one weekend every two weeks in a secondary household).
* Medical clearance from the physician who is treating PCOS.

Exclusion Criteria:

* Physician diagnosis of a major medical illness or eating disorder.
* Fasting blood glucose at or above 126 mg/dL, indicating diabetes mellitus.
* Chronic use of any medication that may affect study outcomes.
* Current smoking.
* Physical, mental, or cognitive handicaps that prevent participation.
* Sister participating in the study.

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Bioavailable Testosterone | Baseline, 6 months

SECONDARY OUTCOMES:
Other Biochemical and Clinical Signs of Hyperandrogenism | Baseline, 6 months
  total and free testosterone, sex hormone binding globulin (SHBG), dehydroepiandrosterone sulfate (DHEAS), hirsutism, acne
Insulin Sensitivity and Beta-cell Function | Baseline, 6 months
  frequently-sampled oral glucose tolerance test, HbA1c
Risk for Cardiovascular Disease | Baseline, 6 months
  serum levels of HDL cholesterol, LDL cholesterol, triglycerides, and C-reactive protein; blood pressure
Body Weight and Composition | Baseline, 6 months
  body fat percentage and distribution assessed by dual-energy x-ray absorptiometry (DXA), waist circumference
Cyclicity of Menstrual Periods | Monthly
Quality of Life | Baseline, 6 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Cara B. Ebbeling, PhD, MS, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ebbeling CB, Leidig MM, Feldman HA, Lovesky MM, Ludwig DS. Effects of a low-glycemic load vs low-fat diet in obese young adults: a randomized trial. JAMA. 2007 May 16;297(19):2092-102. doi: 10.1001/jama.297.19.2092. PMID 17507345
- [Background] Ebbeling CB, Leidig MM, Sinclair KB, Hangen JP, Ludwig DS. A reduced-glycemic load diet in the treatment of adolescent obesity. Arch Pediatr Adolesc Med. 2003 Aug;157(8):773-9. doi: 10.1001/archpedi.157.8.773. PMID 12912783
- [Background] Palmert MR, Gordon CM, Kartashov AI, Legro RS, Emans SJ, Dunaif A. Screening for abnormal glucose tolerance in adolescents with polycystic ovary syndrome. J Clin Endocrinol Metab. 2002 Mar;87(3):1017-23. doi: 10.1210/jcem.87.3.8305. PMID 11889155